CLINICAL TRIAL: NCT02618434
Title: Assessment of the Efficacy and Safety of Molindone Hydrochloride Extended-Release for the Treatment of Impulsive Aggression in Pediatric Patients With Attention Deficit/Hyperactivity Disorder in Conjunction With Standard ADHD Treatment
Brief Title: Treatment of Impulsive Aggression in Subjects With ADHD in Conjunction With Standard ADHD Treatment (CHIME 2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 810P302
Record Dates: First submitted 2015-11-20; First posted 2015-12-01 (Estimated); Results first posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low dose SPN-810 (18 mg) (Experimental): Oral
  Interventions: Drug: SPN-810 (18 mg)
- High dose SPN-810 (36 mg) (Experimental): Oral
  Interventions: Drug: SPN-810 (36 mg)
- Placebo (Placebo Comparator): Oral
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SPN-810 (18 mg) — Subjects were randomized to receive SPN-810 9 mg twice each day with food, in addition to the stable dose of the optimized ADHD medication determined from the lead-in period. If initiating treatment before noon, patients should start with the morning dose; if afternoon, the evening dose.
  Arms: Low dose SPN-810 (18 mg)
Drug: SPN-810 (36 mg) — Subjects were randomized to receive SPN-810 18 mg twice each day with food, in addition to the stable dose of the optimized ADHD medication determined from the lead-in period. If initiating treatment before noon, patients should start with the morning dose; if afternoon, the evening dose.
  Arms: High dose SPN-810 (36 mg)
Drug: Placebo — Subjects were randomized to receive Placebo twice each day with food, in the morning and in the evening, in addition to the stable dose of the optimized ADHD medication determined from the lead-in period. If initiating treatment before noon, patients should start with the morning dose; if afternoon, the evening dose.
  Arms: Placebo

SUMMARY:
The purpose of this study is to demonstrate the efficacy, safety, and tolerability of SPN-810 in the treatment of impulsive aggression in patients with Attention-Deficit/Hyperactivity Disorder (ADHD) in conjunction with standard ADHD treatment. Approximately 297 subjects aged 6 to 12 years with ADHD and comorbid impulsive aggression will be recruited in this study. The frequency of impulsive aggression behaviors will be assessed as a primary outcome. Additionally, the severity and improvement in impulsive aggression and quality of life measures for the subject and caregiver will be assessed using validated scales.

DETAILED DESCRIPTION:
This study is a randomized, placebo-controlled, double-blind, multicenter, parallel group, fixed dose study to demonstrate the efficacy, safety, and tolerability of SPN-810 in the treatment of IA in subjects aged 6 to 12 years with ADHD in conjunction with standard ADHD treatment.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy male or female subjects, age 6 to 12 years at the time of screening with a primary diagnosis of ADHD and currently receiving monotherapy treatment with an optimized FDA-approved ADHD medication.
* Impulsive aggression will be confirmed at screening using R-MOAS and Vitiello Aggression Scale.

Exclusion Criteria:

* Current or lifetime diagnosis of epilepsy, major depressive disorder, bipolar disorder, schizophrenia or a related disorder, personality disorder, Tourette's disorder, or psychosis not otherwise specified.
* Currently meeting DSM criteria for autism spectrum disorder, pervasive developmental disorder, obsessive-compulsive disorder, post-traumatic stress disorder, or any other anxiety disorder as the primary diagnosis.
* Known or suspected intelligence quotient (IQ) < 70, suicidality, pregnancy, or substance or alcohol abuse.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 297 (Actual)
Dates: Start 2016-02-16 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2020-02-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (32):
- United States (32):
  - Metropolitan Neuro Behavioral Institute, Chandler, Arizona
  - Woodland International Research Group, Little Rock, Arkansas
  - Sun Valley Research Center, Imperial, California
  - Alliance for Wellness dba Alliance for Research, Long Beach, California
  - ASCLEPES Research Center, Panorama City, California
  - MCB Clinical Research Centers, LLC, Colorado Springs, Colorado
  - Children's National Medical Center/Children's Research Institute, Washington D.C., District of Columbia
  - Gulfcoast Clinical Research Center, Fort Myers, Florida
  - Indago Research & Health Center, Inc., Hialeah, Florida
  - Innovative Clinical Research, Inc, Lauderhill, Florida
  - Laszlo J. Mate, M.D., P.A., North Palm Beach, Florida
  - APG Research, LLC, Orlando, Florida
  - Miami Research Associates, South Miami, Florida
  - University of South Florida- Dept. of Psychiatry and Neurosciences, Tampa, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - iResearch Atlanta, Decatur, Georgia
  - Advanced Clinical Research, Meridian, Idaho
  - AMR Conventions Research, Naperville, Illinois
  - Pedia Research, Evansville, Indiana
  - Pedia Research, Owensboro, Kentucky
  - Louisiana State University Health Sciences Center, Shreveport, Louisiana
  - St. Charles Psychiatric Associates Midwest Research Center, Saint Charles, Missouri
  - Alivation Research, LLC, Lincoln, Nebraska
  - Quality Clinical Research, Omaha, Nebraska
  - Hassmann Research Institute, Berlin, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of Cincinnati Department of Psychiatry and Behavioral Neuroscience, Cincinnati, Ohio
  - BioBehavioral Research of Austin P.C., Austin, Texas
  - InSite Clinical Research, DeSoto, Texas
  - Houston Clinical Trials, Houston, Texas
  - Ericksen Research & Development, Clinton, Utah
  - Pacific Institute of Medical Sciences, Bothell, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo: Subjects were randomized to receive Placebo twice each day (BID) with food, in the morning and in the evening, in addition to the stable dose of the optimized ADHD medication determined from the lead-in period. If initiating treatment before noon, patients should start with the morning dose; if afternoon, the evening dose.
- Low Dose SPN-810 (18 mg): Oral
  SPN-810 (18 mg): Subjects were randomized to receive SPN-810 9 mg twice each day (BID) with food, in addition to the stable dose of the optimized ADHD medication determined from the lead-in period. If initiating treatment before noon, patients should start with the morning dose; if afternoon, the evening dose.
- High Dose SPN-810 (36 mg): Oral
  SPN-810 (36 mg): Subjects were randomized to receive SPN-810 18 mg twice each day (BID) with food, in addition to the stable dose of the optimized ADHD medication determined from the lead-in period. If initiating treatment before noon, patients should start with the morning dose; if afternoon, the evening dose.
Period: Overall Study
Arm/Group | Placebo | Low Dose SPN-810 (18 mg) | High Dose SPN-810 (36 mg)
Started (The number of subjects is based on the Safety Population which included all randomized subjects who received at least 1 dose of study drug and have at least one post-randomization safety measurements.) | 94 | 56 | 142
Intent-to-Treat (The number of subjects is based on the Intent-to-Treat Population (ITT) which included all subjects who received at least 1 dose of study drug and have a baseline and at least 1 valid post-randomization assessment of frequency of IA behaviors based on IA diary entry.) | 92 | 55 | 140
Modified Intent-to Treat (The number of subjects is based on the Modified Intent-to-Treat Population (mITT) which included all subjects who received at least 1 dose of study drug and had a Baseline IA frequency ≥6 per week and at least 1 valid post-randomization assessment of frequency of IA behaviors based on IA diary entry.) | 90 | 53 | 135
Completed (Safety Population only) | 84 | 45 | 113
Not Completed | 10 | 11 | 29
Not completed — Withdrawal by Subject | 0 | 2 | 3
Not completed — Withdrawal By Parent/Guardian | 5 | 6 | 9
Not completed — Lost to Follow-up | 3 | 1 | 3
Not completed — Adverse Event | 1 | 0 | 12
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Other, Multiple categories | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population: The ITT population includes subjects who received at least one dose of the study drug and have a baseline and at least one valid post-randomization assessment of the frequency of IA behaviors based on an IA diary entry.
Groups:
- Placebo: Subjects treated with a Placebo
- Low Dose SPN-810 (18 mg): Subjects treated with low dose of SPN-810
- High Dose SPN-810 (36 mg): Subjects treated with high dose of SPN-810
- Total: Total of all reporting groups
Arm/Group | Placebo | Low Dose SPN-810 (18 mg) | High Dose SPN-810 (36 mg) | Total
Number analyzed (Participants) | 92 | 55 | 140 | 287
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.3 (1.66) | 9.0 (1.90) | 9.0 (1.87) | 9.1 (1.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 10 | 26 | 56
  Male | 72 | 45 | 114 | 231
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 9 | 24 | 51
  Not Hispanic or Latino | 74 | 45 | 115 | 234
  Unknown or Not Reported | 0 | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 0 | 0 | 2
  Black or African American | 32 | 22 | 44 | 98
  Native Hawaiian or Pacific Islander | 0 | 0 | 1 | 1
  White | 56 | 30 | 91 | 177
  Other | 2 | 3 | 4 | 9
Retrospective-Modified Overt Aggression Scale (R-MOAS) [Mean (Standard Deviation); unit: units on a scale] — R-MOAS scale gauges the severity of aggressive behavior: the frequency of the 16 behaviors is rated over the past week in 4 areas (a-d). For each open question in each area, the parent rates the aggressive behaviors on a scale from 0 to 5 or more times. To each area corresponds a weighted category: 1(a), 4(b), 2(c) and 3(d). Therefore, the sum of each area yields a maximum weighted score of 20 (a), 120 (b), 60 (c), and 90 (c). The total score is the sum of the four area scores or 0-290; the higher the score, the more severe the aggressive behavior is.
  units on a scale | 63.91 (33.430) | 66.38 (27.894) | 67.34 (31.949) | 66.06 (31.637)
Vitiello Aggression Scale [Mean (Standard Deviation); unit: units on a scale] — The Vitiello Aggression Scale is a 10-item rating scale that uses a cluster analysis to categorize aggression into two subtypes; predatory and affective. The predatory score is calculated by summing up the individual scores from items 2, 5, 7, 9, and 10. The affective score is calculated by summing up the individual scores from items 1, 3, 4, 6, and 8. The total score is the difference of predatory score and affective score. Possible range of total score varies from 5 (completely predatory) to -5 (completely affective).
  units on a scale | -3.32 (1.089) | -3.20 (1.129) | -3.48 (1.153) | -3.37 (1.130)

OUTCOME MEASURES:

1. Primary Outcome: Efficacy and Safety of SPN-810 on the Frequency of Impulsive Aggression (IA) Measured by the Impulsive Aggression Diary
Description: The primary efficacy endpoint was percent change (PCHT) in the frequency (unweighted score) of IA behaviors per 7 days in the treatment (titration and maintenance) period relative to the Baseline period calculated over the number of days with non-missing IA diary data. PCHT was then calculated as 100 x (T - B)/B, where T and B are IA behavior frequencies per 7 days during the treatment period (from Day 2 through Visit 6, inclusive) and baseline period (Day ≤1), respectively. The IA behavior frequency per 7 days is defined as (SUM/DAY) x 7, where SUM is the total of the IA behaviors reported in the subject IA diary, and DAY is the number of days with a non-missing IA score in the subject IA diary during the specified study period.
Time Frame: Daily measure from Visit 2 (Week -2) to Visit 6 (Week 5) for a total of 7 weeks
Population: Intent-to-Treat (ITT) Population: The ITT population includes subjects who received at least one dose of the study drug and have a baseline and at least one valid post-randomization assessment of the frequency of IA behaviors based on an IA diary entry. Based on the results of the 810P301 interim analysis, enrollment in the 18 mg of SPN-810 group was halted and subjects planned to receive the 18 mg dose in Stage 2 were randomly assigned to 36 mg of SPN-810 or placebo in a 2:1 ratio.
Measure: Median (Full Range); unit: Percent Change of IA behaviors
Groups:
- High Dose SPN-810 (36 mg): Subjects were randomized to receive SPN-810 18 mg orally twice each day with food, in addition to the stable dose of the optimized ADHD medication determined from the lead-in period. If initiating treatment before noon, patients should start with the morning dose; if afternoon, the evening dose.
Arm/Group | Placebo | High Dose SPN-810 (36 mg)
Number analyzed (Participants) | 90 | 135
Percent Change of IA behaviors | -54.12 [-100.0 to 63.4] | -51.64 [-100.0 to 105.3]
Statistical Analysis 1: Comparison: Placebo vs High Dose SPN-810 (36 mg); Test type: Superiority; p = 0.9383, Wilcoxon (Mann-Whitney); Median Difference (Net) = -0.56, 95% CI 2-sided [-8.96 to 7.84]

2. Secondary Outcome: Effect of SPN-810 on Impulsive Aggression Measured by Clinical Global Impression - Severity Scale (CGI-S)
Description: The Clinical Global Impression - Severity of Illness (CGI-S) is a single item clinician rating of clinician's assessment of the severity of IA behaviors CGI-S was evaluated by the Investigator at each visit on a 7- point scale with 1=Normal, 2=Borderline ill, 3=Mildly ill, 4=Moderately ill, 5=Markedly ill, 6=Severely ill, and 7=Extremely ill. Data represent the change between Baseline (Visit 3/Day 1) and three time points: Visit 4 (Week 1); Visit 5 (Week 2) and Visit 6 (Week 5).
Time Frame: Baseline/Visit 3 (Day 1), Visit 4 (Week 1), Visit 5 (Week 2), and Visit 6 (Week 5). The total duration of the study was 5 weeks.
Population: Intent-to-Treat (ITT) Population: The ITT population included subjects who received at least one dose of the study drug and have a baseline and at least one valid post-randomization assessment of the frequency of IA behaviors based on an IA diary entry.
  Based on the results of the 810P301 interim analysis, enrollment in the 18 mg of SPN-810 group was halted and subjects planned to receive the 18 mg dose in Stage 2 were randomly assigned to 36 mg of SPN-810 or placebo in a 2:1 ratio.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | High Dose SPN-810 (36 mg)
Number analyzed (Participants) | 92 | 140
score on a scale
  Visit 4: number analyzed (Participants) | 91 | 137
  Visit 4 | -0.27 (0.518) | -0.45 (0.776)
  Visit 5: number analyzed (Participants) | 87 | 128
  Visit 5 | -0.67 (0.773) | -0.96 (1.068)
  Visit 6: number analyzed (Participants) | 85 | 111
  Visit 6 | -0.93 (0.997) | -1.06 (1.089)
Statistical Analysis 1: Comparison: Placebo vs High Dose SPN-810 (36 mg); This analysis pertains to Visit 4; Test type: Superiority; p = 0.0979, Mixed Models Analysis; Mean Difference (Net) = -0.15, 95% CI 2-sided [-0.33 to 0.03], Standard Error of Mean 0.090
Statistical Analysis 2: Comparison: Placebo vs High Dose SPN-810 (36 mg); This analysis pertains to Visit 5; Test type: Superiority; p = 0.0502, Mixed Models Analysis; Mean Difference (Net) = -0.25, 95% CI 2-sided [-0.50 to 0.00], Standard Error of Mean 0.126
Statistical Analysis 3: Comparison: Placebo vs High Dose SPN-810 (36 mg); This analysis pertains to Visit 6; Test type: Superiority; p = 0.4769, Mixed Models Analysis; Mean Difference (Net) = -0.10, 95% CI 2-sided [-0.38 to 0.18], Standard Error of Mean 0.141

3. Secondary Outcome: Effect of SPN-810 on Impulsive Aggression Measured by Clinical Global Impression-Improvement (CGI-I) Scale Investigator Rated
Description: The Clinical Global Impression - Improvement Scale (CGI-I) is an assessment of how much the patient's illness has improved or worsened relative to a baseline state at the beginning of treatment.
  CGI-I was evaluated by the Investigator at each visit on a 7-point scale with 1=very much improved, 2= much improved, 3= minimally improved, 4= no change, 5= minimally worse, 6= much worse, 7= very much worse
Time Frame: Visit 4 (Week 1), Visit 5 (Week 2) and Visit 6 (Week 5), a total of 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | High Dose SPN-810 (36 mg)
Number analyzed (Participants) | 92 | 140
score on a scale
  Visit 4: number analyzed (Participants) | 92 | 138
  Visit 4 | 3.4 (0.72) | 3.3 (0.90)
  Visit 5: number analyzed (Participants) | 87 | 129
  Visit 5 | 3.0 (0.97) | 2.7 (0.97)
  Visit 6: number analyzed (Participants) | 85 | 112
  Visit 6 | 2.8 (1.13) | 2.5 (1.04)
Statistical Analysis 1: Comparison: Placebo vs High Dose SPN-810 (36 mg); This analysis pertains to Visit 4; Test type: Superiority; p = 0.0881, Mixed Models Analysis; Mean Difference (Net) = -0.19, 95% CI 2-sided [-0.41 to 0.03], Standard Error of Mean 0.113
Statistical Analysis 2: Comparison: Placebo vs High Dose SPN-810 (36 mg); This analysis pertains to Visit 5; Test type: Superiority; p = 0.0522, Mixed Models Analysis; Mean Difference (Net) = -0.26, 95% CI 2-sided [-0.53 to 0.00], Standard Error of Mean 0.135
Statistical Analysis 3: Comparison: Placebo vs High Dose SPN-810 (36 mg); This analysis pertains to Visit 6; Test type: Superiority; p = 0.1766, Mixed Models Analysis; Mean Difference (Net) = -0.21, 95% CI 2-sided [-0.52 to 0.10], Standard Error of Mean 0.156

4. Secondary Outcome: Effect of SPN-810 on Impulsive Aggression Measured by Child Health Questionnaire Parent Form 28-item (CHQ-PF28)
Description: The CHQ-PF28 is a short generic measure of health status and health-related quality of life. The 28 items have 4, 5, or 6 response options, divided over 8 multi-item scales (physical functioning, general behavior, mental health, self-esteem, general health perceptions, parental impact: emotional, parental impact: time, and family activities) and 5 single item concepts (role functioning: emotional/behavior, role functioning: physical, bodily pain, family cohesion, and change in health). In addition, the individual scale scores will be aggregated to derive 2 summary component scores: the physical functioning and psychosocial health summary scores. The range on subscales and the overall scale is 0-100 (0 = worst possible health state; 100 = best possible health state).
  Data represent the change from Baseline (Visit 3) to one time point, Visit 6 (Week 5).
Time Frame: Baseline Visit 3 (Day 1) and Visit 6 (Week 5). Total duration of the study was 5 weeks.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- High Dose SPN-810 (36 mg): SPN-810 (36 mg): Subjects were randomized to receive SPN-810 18 mg orally twice each day with food, in addition to the stable dose of the optimized ADHD medication determined from the lead-in period. If initiating treatment before noon, patients should start with the morning dose; if afternoon, the evening dose.
Arm/Group | Placebo | High Dose SPN-810 (36 mg)
Number analyzed (Participants) | 92 | 140
score on a scale
  Physical Functioning Summary Score At Visit 6: number analyzed (Participants) | 85 | 112
  Physical Functioning Summary Score At Visit 6 | 7.98 (11.461) | 10.86 (12.120)
  Psychosocial Health Summary Score At Visit 6: number analyzed (Participants) | 85 | 112
  Psychosocial Health Summary Score At Visit 6 | 0.11 (6.150) | -2.29 (9.282)
Statistical Analysis 1: Comparison: Placebo vs High Dose SPN-810 (36 mg); This analysis pertains to the Physical Functioning Summary Score at Visit 6; Test type: Superiority; p = 0.3409, ANCOVA; Mean Difference (Net) = 1.54, 95% CI 2-sided [-1.64 to 4.72], Standard Error of Mean 1.613
Statistical Analysis 2: Comparison: Placebo vs High Dose SPN-810 (36 mg); This analysis pertains to the Psychosocial Health Summary Score at Visit 6; Test type: Superiority; p = 0.0215, ANCOVA; Mean Difference (Net) = -2.21, 95% CI 2-sided [-4.08 to -0.33], Standard Error of Mean 0.952

5. Secondary Outcome: Effect of SPN-810 on Impulsive Aggression Measured by Parenting Stress Index, Fourth Edition, Short Form (PSI-4-SF)
Description: The PSI-4-SF is a 36-item self-report measure of parenting stress. Three subscales Parental Distress (PD), Parent-Child Dysfunctional Interaction (P-CDI), and Difficult Child (DC) consist of 12 items each. Parent chooses one of the 5 responses against each item. The 5 responses are: Strongly Agree (SA), Agree (A), Not Sure (NS), Disagree (D), and Strongly Disagree (SD) to indicate the degree to which they agree with each statement. The PD subscale raw score ranges from 12-60, P-CDI and DC each subscale raw score ranges from 16-56. The total stress raw score is the sum of the three subscales (PD+P-CDI+ DC) with a minimum score of 44 and a maximum score of 172. The total stress score is then converted into the percentile score. Parents with a 91st percentile or higher are experiencing clinically significant levels of stress. Data represents the mean change in percentile score from Baseline (Visit 3) and one time point, Visit 6 (Week 5).
Time Frame: Baseline Visit 3 (Day 1) and Visit 6 (Week 5). Total duration of the study was 5 weeks.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | High Dose SPN-810 (36 mg)
Number analyzed (Participants) | 92 | 140
score on a scale
  Total Score at Visit 6: number analyzed (Participants) | 85 | 107
  Total Score at Visit 6 | -5.29 (12.830) | -7.38 (15.757)
  Parental Distress Domain at Visit 6: number analyzed (Participants) | 85 | 109
  Parental Distress Domain at Visit 6 | -1.02 (5.486) | -1.05 (6.313)
  Parent-Child Dysfunctional Interaction Domain at Visit 6: number analyzed (Participants) | 85 | 107
  Parent-Child Dysfunctional Interaction Domain at Visit 6 | -2.13 (5.593) | -2.42 (6.663)
  Difficult Child Domain at Visit 6: number analyzed (Participants) | 85 | 109
  Difficult Child Domain at Visit 6 | -2.14 (5.898) | -3.94 (6.406)
Statistical Analysis 1: Comparison: Placebo vs High Dose SPN-810 (36 mg); This analysis pertains to the Total Score at Visit 6; Test type: Superiority; p = 0.5977, ANCOVA; Mean Difference (Net) = -1.06, 95% CI 2-sided [-5.00 to 2.89], Standard Error of Mean 2.000
Statistical Analysis 2: Comparison: Placebo vs High Dose SPN-810 (36 mg); This analysis pertains to the Parental Distress Domain score at Visit 6; Test type: Superiority; p = 0.8049, ANCOVA; Mean Difference (Net) = 0.20, 95% CI 2-sided [-1.39 to 1.79], Standard Error of Mean 0.807
Statistical Analysis 3: Comparison: Placebo vs High Dose SPN-810 (36 mg); This analysis pertains to the Parent-Child Dysfunctional Interaction score at Visit 6; Test type: Superiority; p = 0.8911, ANCOVA; Mean Difference (Net) = 0.11, 95% CI 2-sided [-1.47 to 1.69], Standard Error of Mean 0.801
Statistical Analysis 4: Comparison: Placebo vs High Dose SPN-810 (36 mg); This analysis pertains to the Difficult Child Domain score Visit 6; Test type: Superiority; p = 0.1426, ANCOVA; Mean Difference (Net) = -1.25, 95% CI 2-sided [-2.93 to 0.42], Standard Error of Mean 0.849

6. Secondary Outcome: Effect of SPN-810 on Impulsive Aggression Measured by Clinical Global Impression-Improvement (CGI-I) Scale Caregiver Rated
Description: The CGI scale was developed to provide a brief, stand-alone assessment of the clinician's view of a subjects' global functioning prior to and after administration of a study medication. The scale was also rated by the Caregiver to assess the improvement of IA behaviors.
  . CGI-I was evaluated by the Caregiver at each visit on a 7-point scale with 1=very much improved, 2= much improved, 3= minimally improved, 4= no change, 5= minimally worse, 6= much worse, 7= very much worse
Time Frame: Visit 4 (Week 1), Visit 5 (Week 2) and Visit 6 (Week 5), a total of 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | High Dose SPN-810 (36 mg)
Number analyzed (Participants) | 92 | 140
score on a scale
  Visit 4 | 3.1 (0.95) | 3.1 (1.02)
  Visit 5 | 2.9 (1.14) | 2.7 (0.94)
  Visit 6 | 2.7 (1.26) | 2.5 (1.12)
Statistical Analysis 1: Comparison: Placebo vs High Dose SPN-810 (36 mg); This analysis pertains to Visit 4; Test type: Superiority; p = 0.6171, Mixed Models Analysis; Mean Difference (Net) = -0.07, 95% CI 2-sided [-0.33 to 0.20], Standard Error of Mean 0.134
Statistical Analysis 2: Comparison: Placebo vs High Dose SPN-810 (36 mg); This analysis pertains to Visit 5; Test type: Superiority; p = 0.0617, Mixed Models Analysis; Mean Difference (Net) = -0.27, 95% CI 2-sided [-0.55 to 0.01], Standard Error of Mean 0.143
Statistical Analysis 3: Comparison: Placebo vs High Dose SPN-810 (36 mg); This analysis pertains to Visit 6; Test type: Superiority; p = 0.4419, Mixed Models Analysis; Mean Difference (Net) = -0.13, 95% CI 2-sided [-0.47 to 0.21], Standard Error of Mean 0.171

7. Secondary Outcome: Effect of SPN-810 on Impulsive Aggression Measured by the Swanson, Nolan, Pelham Rating Scale- Revised (SNAP-IV) Rating Scale
Description: The Swanson, Nolan, Pelham Rating Scale-Revised (SNAP-IV) includes 18 ADHD and 8 oppositional defiant disorder (ODD) symptoms. The symptoms are scored on a 4-point scale, not at all=0, just a little=1, Quite a bit= 2, very much=3. The ratings from the SNAP-IV scale are grouped into the following 4 subscales: ADHD Inattention (items #1-9), ADHD Hyperactivity/Impulsivity (items#10-18), ODD (items# 19-26), and ADHD-combined (first two scales combined, items #1-18). Each observed subscale score is the average rating of the items scores for the subscale where scores range from 0-3; the higher is the score, worsen is the outcome.
  Data represent the change of the observed scores between Baseline (Visit 3) and the end of the study, Visit 6 (Week 5).
Time Frame: Baseline Visit 3 (Day 1) and Visit 6 (Week 5). Total duration of the study was 5 weeks.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | High Dose SPN-810 (36 mg)
Number analyzed (Participants) | 92 | 140
score on a scale
  Inattention subscale: number analyzed (Participants) | 85 | 112
  Inattention subscale | -0.33 (0.539) | -0.46 (0.593)
  Hyperactivity/Impulsivity subscale: number analyzed (Participants) | 85 | 112
  Hyperactivity/Impulsivity subscale | -0.33 (0.590) | -0.50 (0.681)
  Oppositional Defiant Disorder subscale: number analyzed (Participants) | 85 | 112
  Oppositional Defiant Disorder subscale | -0.50 (0.685) | -0.60 (0.732)
  Combined subscale: number analyzed (Participants) | 85 | 112
  Combined subscale | -0.33 (0.501) | -0.48 (0.576)
Statistical Analysis 1: Comparison: Placebo vs High Dose SPN-810 (36 mg); This analysis pertains to the Inattention subscale at Visit 6; Test type: Superiority; p = 0.0416, ANCOVA; Mean Difference (Net) = -0.16, 95% CI 2-sided [-0.32 to -0.01], Standard Error of Mean 0.080
Statistical Analysis 2: Comparison: Placebo vs High Dose SPN-810 (36 mg); This analysis pertains to Hyperactivity/Impulsivity subscale at Visit 6; Test type: Superiority; p = 0.0921, ANCOVA; Mean Difference (Net) = -0.15, 95% CI 2-sided [-0.33 to 0.02], Standard Error of Mean 0.089
Statistical Analysis 3: Comparison: Placebo vs High Dose SPN-810 (36 mg); This analysis pertains to the Oppositional Defiant Disorder subscale at Visit 6; Test type: Superiority; p = 0.4480, ANCOVA; Mean Difference (Net) = -0.07, 95% CI 2-sided [-0.26 to 0.11], Standard Error of Mean 0.094
Statistical Analysis 4: Comparison: Placebo vs High Dose SPN-810 (36 mg); This analysis pertains to the Combined Scale score at Visit 6; Test type: Superiority; p = 0.0457, ANCOVA; Mean Difference (Net) = -0.16, 95% CI 2-sided [-0.31 to -0.00], Standard Error of Mean 0.077

8. Secondary Outcome: Effect of SPN-810 on Impulsive Aggression Measured by the Percentage of Responders
Description: A Responder was defined as a subject with at least a 30% or 50% reduction in the frequency of IA behaviors per 7 days in the Treatment (Titration and Maintenance) period relative to the Baseline period per the IA Diary.
  Data represent the percentage of subjects with 30% and 50% reduction in IA behaviors from Baseline to end of treatment period.
Time Frame: Daily measure from Visit 2 (Week -2) to Visit 6 (Week 5) for a total of 7 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo | High Dose SPN-810 (36 mg)
Number analyzed (Participants) | 92 | 140
percentage of subjects
  ≥ 30% Responder | 73.9 | 75.0
  ≥ 50% Responder | 54.3 | 51.4
Statistical Analysis 1: Comparison: Placebo vs High Dose SPN-810 (36 mg); This analysis pertains to ≥ 30% Responders; Test type: Superiority; p = 0.8525, Regression, Logistic; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.58 to 1.93]
Statistical Analysis 2: Comparison: Placebo vs High Dose SPN-810 (36 mg); This analysis pertains to ≥ 50% Responders; Test type: Superiority; p = 0.6635, Regression, Logistic; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.52 to 1.51]

ADVERSE EVENTS:
Time Frame: Visit 3 (Day 1) to Visit 7 (Week 6)-End of Study, a total of 6 weeks
Description: Adverse events reporting pertains to the Safety Population which include all randomized subjects who received at least 1 dose of study drug and have at least one post-randomization safety measurements.
Groups:
- Low Dose SPN-810 (18 mg): Subjects were randomized to receive SPN-810 9 mg orally twice each day with food, in addition to the stable dose of the optimized ADHD medication determined from the lead-in period. If initiating treatment before noon, patients should start with the morning dose; if afternoon, the evening dose.
Arm/Group | Placebo | Low Dose SPN-810 (18 mg) | High Dose SPN-810 (36 mg)
All-Cause Mortality (participants affected / at risk) | 0/94 | 0/56 | 0/142
Serious Adverse Events (participants affected / at risk) | 1/94 | 0/56 | 4/142
Other Adverse Events (participants affected / at risk) | 13/94 | 10/56 | 23/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=94) | Low Dose SPN-810 (18 mg) (N=56) | High Dose SPN-810 (36 mg) (N=142)
Post-Traumatic Stress Disorder (Psychiatric disorders) | 1 | 0 | 0
Drug Hypersensitivity (Immune system disorders) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 1
Dystonia (Nervous system disorders) | 0 | 0 | 1
Aggression (Psychiatric disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=94) | Low Dose SPN-810 (18 mg) (N=56) | High Dose SPN-810 (36 mg) (N=142)
Headache (Nervous system disorders) | 8 | 3 | 14
Vomiting (Gastrointestinal disorders) | 3 | 4 | 6
Blood prolactin increase (Investigations) | 2 | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-03-29): https://cdn.clinicaltrials.gov/large-docs/34/NCT02618434/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-21): https://cdn.clinicaltrials.gov/large-docs/34/NCT02618434/SAP_001.pdf